CLINICAL TRIAL: NCT01602406
Title: A Multicenter, Open-label, Dose Escalation, Phase I Study of LJM716 Administered Intravenously in Combination With Trastuzumab in Patients With HER2 Overexpressing Metastatic Breast Cancer or Gastric Cancer
Brief Title: Phase I Study LJM716 Combined With Trastuzumab in Patients With HER2 Overexpressing Metastatic Breast or Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLJM716X2102; 2011-004881-13 (EudraCT Number)
Record Dates: First submitted 2012-05-07; First posted 2012-05-21 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2018-07

CONDITIONS: Advanced HER2-positive Breast Cancer or Gastric Cancer
Keywords: Advanced HER2-positive Breast cancer or Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — elgemtumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LJM716 in combination with trastuzumab (Experimental)
  Interventions: Drug: LJM716; Drug: Trastuzumab

INTERVENTIONS:
Drug: LJM716 — LJM716
Drug: Trastuzumab — Trastuzumab

SUMMARY:
This is a multicenter, open-label, dose escalation, phase I study to estimate the Maximum Tolerated Dose (MTD) or a lower Recommended Dose for Expansion (RDE) of LJM716 in combination with trastuzumab in patients with Human Epidermal growth factor Receptor 2 (HER2) overexpressing Metastatic Breast Cancer (MBC) or gastric cancer (MGC). The study consists of a dose escalation part and a dose expansion part. LJM716 will be administered intravenously once weekly unless a less frequent dosing regimen such as every 2 weeks or once every 4 weeks is introduced. Patients will continue on their trastuzumab dosing, administered intravenously once weekly at 2mg/kg. During dose escalation, a minimum of 15 patients are anticipated to be treated in successive cohorts. The dose escalation will continue until the MTD/RDE is declared. The RDE dose selected will either be the MTD or a dose below the MTD based on safety and Pharmacokinetic/Pharmacodynamic (PK/PD) considerations. Following the MTD/RDE declaration, approximately 20 MBC and 20 MGC patients will be enrolled in separate arms in the dose expansion part and treated at the MTD/RDE to further assess the safety, tolerability, and anti-tumor activity of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed HER-2 positive, metastatic or non-operable locally advanced breast or gastric cancer
* Metastatic breast cancer patients must have received a minimum of 1 and a maximum of 3 prior anti HER2 based regimens with documented progression on the most recent regimen which must contain trastuzumab, ado-trastuzumab emtansine or lapatinib
* Metastatic gastric cancer patients must have received a minimum of 1 and a maximum of 2 prior anti HER2 based regimens with documented progression on the most recent regimen which must contain trastuzumab or ado-trastuzumab emtansine
* During the dose expansion part of study, all patients must have at least one measurable lesion as defined by RECIST criteria.
* Patients must have at least one prior trastuzumab-containing regimen
* Eastern Cooperative Oncology Group (ECOG) Performance status ≤ 2

Exclusion Criteria:

* Patients with Central Nervous System (CNS) metastasis which are: symptomatic or require treatment for symptom control and/or growing
* Prior treatment with any anti-HER3 (Human Epidermal growth factor Receptor 3) treatment
* Impaired cardiac function
* Prior to the first dose of study treatment, patients who have received systemic antineoplastic therapy or any investigational therapy within 4 weeks or within 5 half- lives of the therapy prior to starting study treatment, whichever is shorter, or for cyclical therapy, within one cycle length (e.g. 6 weeks for nitrosourea, mitomycin-C).
* Patients who have a history of primary malignancy other than that being treated in this study, and currently requires active clinical intervention.
* Patients who do not have an archival tumor sample (or sections of it) available or readily obtainable.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-09-21 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Incidence rate of Dose Limiting Toxicities | 4 weeks
  Incidence of dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Number of adverse events | 4 months
  Safety assessment
Number of serious adverse events | 4 months
  Safety assessment
Pharmacodynamic response to LJM716 in tumor tissue | 3 months
  Post-treatment change from baseline in pHER3 levels in the tumor
Progression-free survival | 18 months
  Efficacy assessment
Duration of response | 18 months
  Efficacy assessment
Serum concentration of anti-LJM716 antibodies | 4 months
  Incidence of antibodies against LJM716
Serum concentration of LJM716 when administered in combination with trastuzumab | 4 months
  PK profile
Frequency of partial responses according to Response Evaluation Criteria In Solid Tumors (RECIST) | every 2 months up to 18 months
  Efficacy assessment
Frequency of complete responses according to RECIST | every 2 months up to 18 months
  Efficacy assessment
Frequency of stable disease according to RECIST | every 2 months up to 18 months
  Efficacy assessment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (3):
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Philadelphia, Pennsylvania
- Novartis Investigative Site, Wilrijk, Belgium
- Novartis Investigative Site, Saint-Herblain, France
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Seoul, Korea, South Korea
- Novartis Investigative Site, Valencia, Valencia, Spain
- Novartis Investigative Site, Taipei, Taiwan
- Novartis Investigative Site, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLJM716X2102 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17162